CLINICAL TRIAL: NCT05308693
Title: Evaluation of the Effect of Two Different Methods in Teaching Stoma Care Skills in Patients With Stoma on Stoma Compliance and Self-efficacy Level of Patients
Brief Title: Evaluation of the Effect of Two Different Methods on Stoma Compliance and Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Acibadem University, Asisst. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2021-13/04
Record Dates: First submitted 2022-03-03; First posted 2022-04-04 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Patient Relations, Nurse; Patient Satisfaction
Keywords: Stoma Adaptation; Self efficacy; Stoma Care education
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-Classical patient education (No Intervention): Before the operation, the stoma area is marked, the patient is educated with the classical method brochure
- Experimental-Patient Compatible Stoma Educational Material (Experimental): The stoma area is marked before the operation; A brochure is given to the patient. Practical training is given on the patient's own body with patient-compatible stoma training material.
  Interventions: Other: Education material - Patient Compatible Stoma Educational Material

INTERVENTIONS:
Other: Education material - Patient Compatible Stoma Educational Material — It is an educational material made of rubber, similar to a stoma, that can be placed on the patient.
  Arms: Experimental-Patient Compatible Stoma Educational Material

SUMMARY:
In patients with stoma, apart from traditional methods, different methods whşch can be used in visual, auditory and motor skills are recommended as a part of education methods regarding stoma care.

The aim of this study is to evaluate the effects of two different methods in teaching stoma care skills considering patients with colostomy/ileostomy on stoma compliance and self-efficacy levels. This research is the thesis study designed within the scope of the Surgical Diseases Nursing Master's program.

DETAILED DESCRIPTION:
Stoma is the opening of the intestine to the abdominal wall. In recent years, the number of individuals with ostomy has been increasing, and it is stated that there are 800,000 individuals in North America alone and approximately 15,000 in Hong Kong.. As a result of this surgical procedure, regardless of ileostomy or colostomy, the daily life of individuals who went through this procedure has been affected in terms of not only the way their bodies excretes but also way of their eating habits, sexual life, self-esteem, religious/cultural needs, social life, sense of independence, self-care and the rest of their daily life.. Gaining patients' self-care activities related to stoma care begins in the preoperative period.

The self-care and development of activities in patients with stoma consists of cognitive, emotional, and psychomotor learning processes.

Patients need to acquire the necessary knowledge and skills to meet their new care needs. This learning process is based on the nurse's practical experience and teaching methods.. After the surgery of individuals with stoma; these individuals need training and counseling in order to manage the stoma functionally and to adapt a life with a stoma in psychological terms. Wound ostomy incontinence nurses; are an unique source of information when it comes to educating the individuals who have stoma.. The American Society of Colon and Rectal Surgeons recommends preoperative stoma training. In the post-operative period after a proper training given to individuals with stoma; It is stated that reduces stoma-related complications, shortens hospital stay, and reduces the cost of stoma care. In the literature, it is stated that the stoma training performed before the surgery shortens the discharge time, reduces the cost and improves the adequacy of the individuals.. The environment, duration, patient's readiness level, past knowledge and experience of patient, education method to be used, education content and material have an important place in patient training. The language of instruction should be plain and simple.. Today, in patient training, verbal information is provided by giving written materials or showing the care practices on the patient after the surgery. While increasing the permanence and effectiveness of the materials used with the developing technology, educational content such as brochures, models, booklets, question-answers, videos and slides also provide good results. However, since the socio demographic characteristics and learning styles of the patients are different from each other, the desired permanence may not be fully achieved. Since stoma care is frequently encountered in nursing practices, is of vital importance, and affects the quality of health care of the individual, family and society, overall it is expected that the permanence of education in this practice will be increased using audio-visual and motor skills, behavior change and self-efficacy will be improved considering the increasing compliance situation in patients with stoma.. Pouresmail et al. (2019) shows that the use of simulation to learn ostomy self-care improves self-efficacy in patients.. In the literature, studies on the subject are limited, and the aim of this study is to determine the effects of two different methods in stoma care education on stoma compliance and self-efficacy levels of patient

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-85 years
* Patients who have a colostomy or ileostomy for any reason (cancer, ulcerative colitis, chron, hernia, etc.)
* Patients who can speak and understand Turkish and do not have a psychological or neurological disease (Advanced Parkinson's, Alzheimer's, Depression, etc.)

Exclusion Criteria:

* Patients with visual and hearing impairment
* Patients that are unable to use their hands and upper extremities (hemiplegic, paraplegic, etc.)
* Patients who requires a revision surgery after surgery
* Patients whose temporary stoma was closed while in the data collection process
* Patients with postoperative complications and prolonged discharge period (evisceration, bleeding, perforation, etc.) will be excluded from the sample.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
State Anxiety Level | after surgery, post-operative 1. day (first stoma care)
  State Anxiety Level is evaluated by Spielberger State-Trait Anxiety Inventory - This inventory is a four-degree Likert type scale ranging from "Almost never" to "Almost always". In the state anxiety scale, the individual evaluates how he/ she feels "right now". The total score obtained from each scale varies between 20 and 80. A high score indicates a high anxiety level, a low score indicates a low anxiety level

SECONDARY OUTCOMES:
Stoma Self-Efficacy Scale | The scale is filled in 3 times; 3 days after the surgery (post-operative 3. day) in hospital (1), and at the 3rd week after surgery (post-operative 21. day) at home by telephone (2) and 9th week after surgery (post-operative 63. day) (3) at home by phone
  In order to determine the self-efficacy levels of individuals with stoma, the psychometric properties of the scale were examined in English, Knippenberg, Van Berge-Henegouwen in 1996. Turkish validity and reliability of the scale Karaçay et al. Adapted by (2020). The scale consists of 22 items. The scale, which is graded in a five-point Likert type, consists of two sub-dimensions. Sub-dimensions; Stoma Care is Self-Efficacy and Social Self-Efficac. The possible score on the scale ranges from 22 to 110. The higher the score, the better the level of self-efficacy

OTHER OUTCOMES:
Adjustment Scale for Individuals with Ostomy | The scale is filled in 3 times; 3 days after the surgery (post-operative 3. day) in hospital (1), and at the 3rd week after surgery (post-operative 21. day) at home by telephone (2) and 9th week after surgery (post-operative 63. day) (3) at home by phone
  It is a self-assessment scale consisting of 23 items developed by Simmsons, Smith, and Maekawa to determine the compliance of individuals with stoma. Adjustment Scale for Individuals with Ostomy Karadağ et al. (2011), adapted into Turkish. The scale, which is graded in a five-point Likert type, has four sub-dimensions. These four dimensions are anger, social adaptation, anxiety/worry and acceptance. While the lowest score on the scale is '0', the highest score is '92'.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Uslu, Asisst.Prof, Study Director — Acıbadem Mehmet Ali Aydınlar Üniversitesi
Locations (1):
- Yasemin Uslu, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karacay P, Togluk Yigitoglu E, Karadag A. The validity and reliability of the Stoma Self-Efficacy Scale: A methodological study. Int J Nurs Pract. 2020 Dec;26(6):e12840. doi: 10.1111/ijn.12840. Epub 2020 Apr 17. PMID 32301580
- [Result] Stelton S. CE: Stoma and Peristomal Skin Care: A Clinical Review. Am J Nurs. 2019 Jun;119(6):38-45. doi: 10.1097/01.NAJ.0000559781.86311.64. PMID 31135430
- [Result] Giordano V, Nicolotti M, Corvese F, Vellone E, Alvaro R, Villa G. Describing self-care and its associated variables in ostomy patients. J Adv Nurs. 2020 Nov;76(11):2982-2992. doi: 10.1111/jan.14499. Epub 2020 Aug 26. PMID 32844474
- [Result] Seo HW. Effects of the frequency of ostomy management reinforcement education on self-care knowledge, self-efficacy, and ability of stoma appliance change among Korean hospitalised ostomates. Int Wound J. 2019 Mar;16 Suppl 1(Suppl 1):21-28. doi: 10.1111/iwj.13047. PMID 30793857
- [Result] Zhang Y, Xian H, Yang Y, Zhang X, Wang X. Relationship between psychosocial adaptation and health-related quality of life of patients with stoma: A descriptive, cross-sectional study. J Clin Nurs. 2019 Aug;28(15-16):2880-2888. doi: 10.1111/jocn.14876. Epub 2019 May 5. PMID 30939212
- [Result] Cheng F, Meng AF, Yang LF, Zhang YN. The correlation between ostomy knowledge and self-care ability with psychosocial adjustment in Chinese patients with a permanent colostomy: a descriptive study . Ostomy Wound Manage. 2013 Jul;59(7):35-8. PMID 23846005